CLINICAL TRIAL: NCT04783116
Title: The Effects of Plant Stanol Ester Supplements on Liver Inflammation in Overweight and Obese Children
Brief Title: Plant Stanols and Liver Inflammation in Overweight and Obese Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL73527.000.20
Record Dates: First submitted 2021-02-23; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; NAFLD; NASH; NASH - Nonalcoholic Steatohepatitis; Childhood Obesity; Childhood Overweight; Pediatric Obesity
Keywords: Non-alcoholic Fatty Liver Disease; NAFLD; NASH; Non-alcoholic Steatohepatitis; Liver inflammation; Overweight; Obesity; Adolescents; Children; Lifestyle; Combined lifestyle intervention
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity; Hepatitis; Overweight; Obesity | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant stanols (3g/day) (Experimental): Consumption of plant stanol chews
  Interventions: Dietary Supplement: Plant stanols (3g/day)
- Control (Placebo Comparator): Consumption of placebo chews (without plant stanols)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plant stanols (3g/day) — Oral consumption of 6 plant stanol enriched chews per day for 6 months (total dosage is 3g/day). Chews are consumed with main meals: two with breakfast, two with lunch and two with dinner.
  Other Names: Benecol (Raisio Nutrition Ltd., Raisio, Finland)
  Arms: Plant stanols (3g/day)
Dietary Supplement: Placebo — Oral consumption of 6 placebo chews per day for 6 months. Chews are consumed with main meals: two with breakfast, two with lunch and two with dinner.
  Arms: Control

SUMMARY:
Obesity is associated with a variety of co-morbidities. Children with obesity are more likely to have risk factors associated with cardiovascular diseases (CVD) and CVD risk markers (e.g. hypertension, elevated serum cholesterol, and type 2 diabetes mellitus), but also with organ specific pathologies such as a non-alcoholic fatty liver disease (NAFLD). A recent meta-analysis has shown that the prevalence of NAFLD in obese pediatric populations is approximately 35%, compared to approximately 8% in general pediatric population, making it a very important health threat in these populations. Successful pharmacological interventions to treat or prevent NASH are not yet available and so far only weight loss has clear benefits. However, it is well known that sustained weight-loss is difficult to achieve on the longer-term. The investigators recently demonstrated in mice that plant sterol and stanol ester consumption inhibited the development of liver inflammation. Moreover, Javanmardi et al. recently demonstrated in a population of adult NAFLD patients, that plasma concentrations of Alanine Transaminase (ALT) were reduced after daily plant sterol consumption (1.6 g/d) for 6 weeks. In this study, the investigators propose to evaluate the effect of consuming soft chews enriched with plant stanol esters (3 grams/day) on ALT concentrations in children with overweight or (morbid) obesity who are at risk of developing NAFLD, in a randomized, placebo-controlled, double blinded study with an intervention period and follow-up period of 6 months. 52 overweight and obese children with elevated ALT concentrations (>39 U/L for boys and >33 U/L for girls) will be included. All children will be randomly allocated to consume control or plant stanol ester enriched soft chews on a daily basis for a period of 6 months. After 12 months there will be an additional blood sample to evaluate whether the 6 months intervention is still effective.

ELIGIBILITY:
Inclusion Criteria:

* Participation in lifestyle intervention, provided by the Centre for Overweight Adolescent and Children Healthcare (COACH), at the Department of Pediatrics at the Maastricht University Medical Center (MUMC+).
* Age between 4-18 years old
* Plasma ALT concentrations above 39 U/L for boys and above 33 U/L for girls.
* Willingness to consume 6 soft chews on a daily basis, for a period of 6 months.

Exclusion Criteria:

* Presence of a severe medical condition, which contraindicates, in the investigators judgement, entry to the study.
* No signed informed consent by relevant parties (parents of children aged below 12 years, parents and or children aged between 12 and 16 years, or children aged 16 years and older).

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma ALT concentration at 6 and 12 months. | Baseline, 6 months and 12 months
  Plasma ALT (Alanine Aminotransferase) concentration is a laboratory parameter, measured in blood, reflecting possible presence of NAFLD. Concentrations below 26 U/L for boys, and below 22 U/L for girls, are considered normal. Concentrations above 39 U/L for boys, and above 33 U/L are considered to reflect presence of NAFLD.

SECONDARY OUTCOMES:
Change in plasma AST and plasma CK-18 concentration at 6 and 12 months. | Baseline, 6 months and 12 months
  Aspartate Aminotransferase (AST) and cytokeratin-18 (CK-18) are laboratory parameters, measured in the participants blood in U/L, reflecting liver health.
Change in liver inflammation parameters at 6 and 12 months. | Baseline, 6 months and 12 months
  Cathepsin-D and acid phosphatase are laboratory parameters, measured in mg/L in the participants blood, reflecting liver inflammation.
Change in lipid metabolism parameters at 6 and 12 months. | Baseline, 6 months and 12 months
  Serum total cholesterol, HDL cholesterol, triacylglycerol (TAG) with correction for free glycerol and non-esterified fatty acids (NEFA) are laboratory parameters, measured in mmol/L in the participants blood, reflecting their lipid metabolism.
Change in lipid protein metabolism parameters at 6 and 12 months. | Baseline, 6 months and 12 months
  ApoA1 and apoB100 plasma concentrations are laboratory parameters, measured in g/L in the participants blood, reflective of the lipoprotein metabolism.
Change in plasma glucose concentration at 6 and 12 months. | Baseline, 6 months and 12 months
  Fasting glucose is a laboratory parameter, measured in mmol/L in the participants blood, reflecting glucose metabolism.
Change in plasma insulin concentration at 6 and 12 months. | Baseline, 6 months and 12 months
  Fasting insulin concentrations is a laboratory parameters, measured in mU/L in the participants blood, reflecting glucose metabolism.
Change in insulin sensitivity at 6 and 12 months. | Baseline, 6 months and 12 months
  Insulin sensitivity will be calculated using the HOMA-IR formula (homeostatis model) which is (fasting glucose*fasting insulin) /22,5. As HOMA-IR is a ratio, it does not have a unit.
Change in non-cholesterol sterol and oxy(phyto)sterol concentrations at 6 and 12 months. | Baseline, 6 months and 12 months
  A panel of non-cholesterol sterols, as surrogate markers for cholesterol absorption and synthesis will be measured in the participants blood.
Change in plasma inflammatory markers at 6 and 12 months. | Baseline, 6 months and 12 months
  Plasma concentrations of CRP and high sensitivity CRP will be measured in mg/L in the participants blood, to assess presence of low-grade inflammation in the body.
Change in ultrasonographic hepatorenal index (HRI) at 6 and 12 months. | Baseline, 6 months and 12 months
  HRI is measured during a conventional ultrasound of the liver, in which three close-up images of the liver and right kidney are made by a physician-researcher. HRI is calculated from these images by a pediatric radiologist, as the ratio of the hepatic brightness and the renal brightness (HRI = echogenicity of the liver/echogenicity of the kidney). The average of the three images is taken as the definite HRI, as a reflection of hepatic fat content.
Change in continuous Controlled Attenuation Parameter (CAP) at 6 and 12 months. | Baseline, 6 months and 12 months
  CAP is measured during a vibration controlled transient elastography of the liver, which is performed with a Fibroscan by a physician-researcher. The value is a reflection of hepatic fat content.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No